CLINICAL TRIAL: NCT05279014
Title: The Effect of Fasted Exercise on LDL-cholesterol in Men and Women
Brief Title: Fasted Exercise and LDL-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: King's College London (Other); Zoe Global Limited (Other)
Responsible Party: Principal Investigator, Louise Bradshaw, PhD Student, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EIRA1-7137
Record Dates: First submitted 2022-02-16; First posted 2022-03-15 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise in a fed-state (Active Comparator): 12-weeks of exercise training, 50-minutes, 3 days per week performed 1.5-3 hours after a high-carbohydrate meal (1 g/kg body mass).
  Interventions: Other: Meal timing
- Exercise in a fasted-state (Experimental): 12-weeks of exercise training, 50-minutes, 3 days per week performed after at least an 8-hour fast. A high-carbohydrate meal (1 g/kg body mass) will be consumed after exercise.
  Interventions: Other: Meal timing

INTERVENTIONS:
Other: Meal timing — A high-carbohydrate (1 g/kg body mass) meal to be consumed either 1.5-3 hours before or immediately after exercise. Those consuming the meal after exercise will have fasted for at least 8 hours before exercise.

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in the UK and worldwide with low density lipoprotein cholesterol (LDL-C) being one of the most important modifiable risk factors. Physical activity is inexpensive and research shows that it consistently improves high density lipoprotein and triglyceride concentrations. However, fails to improve LDL-C concentrations. Preliminary research suggests fasted exercise could potentially improve LDL-C concentrations. The majority of research in these areas have also mostly been done in males with the results generalised to females. As it is known that lipid metabolism and CVD risk is different between sexes it is possible that the response to fasted exercise may also be different between sexes. This aim of this study is to assess the effect of physical activity performed before or after a meal on plasma LDL-C concentrations in men and women and explore sex differences. The study will also assess the effect of fasted exercise on other CVD risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Body mass index 20-40kg/m2
* Physically inactive (exercise for less than 150 minutes per week)

Exclusion Criteria:

* Weight instability (>5kg change in body mass over last 6 months)
* Diagnosis of diabetes or CVD
* Pregnant or lactating
* Any medical condition or medication that could introduce bias into the study (eg. lipid disorders, lipid or glucose metabolism altering medications eg statins)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Change in fasting plasma LDL-C concentrations at week 12 | Baseline and week 12
  Fasting plasma LDL-cholesterol concentrations (mmol/L)

SECONDARY OUTCOMES:
Change in fasting plasma LDL-C concentrations at week 4 | Baseline and week 4
  Fasting plasma LDL-cholesterol concentrations (mmol/L)
Change in fasting plasma HDL-C concentrations at week 12 | Baseline and week 12
  Fasting plasma HDL-cholesterol concentrations (mmol/L)
Change in fasting plasma HDL-C concentrations at week 4 | Baseline and week 4
  Fasting plasma HDL-cholesterol concentrations (mmol/L)
Change in fasting plasma total cholesterol concentrations at week 12 | Baseline and week 12
  Fasting plasma total cholesterol concentrations (mmol/L)
Change in fasting plasma total cholesterol concentrations at week 4 | Baseline and week 4
  Fasting plasma total cholesterol concentrations (mmol/L)
Change in fasting plasma apolipoprotein B concentrations at week 12 | Baseline and week 12
  Fasting plasma apolipoprotein B concentrations (mmol/L)
Change in fasting plasma apolipoprotein B concentrations at week 4 | Baseline and week 4
  Fasting plasma apolipoprotein B concentrations (mmol/L)
Change in fasting plasma triglyceride concentrations at week 12 | Baseline and week 12
  Fasting plasma triglyceride concentrations (mmol/L)
Change in fasting plasma triglyceride concentrations at week 4 | Baseline and week 4
  Fasting plasma triglyceride concentrations (mmol/L)
Change in fasting plasma C-reactive protein concentrations at week 12 | Baseline and week 12
  Fasting plasma C-reactive protein concentrations (mg/L)
Change in fasting plasma C-reactive protein concentrations at week 4 | Baseline and week 4
  Fasting plasma C-reactive protein concentrations (mg/L)
Change in fasting plasma glucose concentrations at week 12 | Baseline and week 12
  Fasting plasma glucose concentrations (mmol/L)
Change in fasting plasma glucose concentrations at week 4 | Baseline and week 4
  Fasting plasma glucose concentrations (mmol/L)
Change in fasting plasma insulin concentrations at week 12 | Baseline and week 12
  Fasting plasma insulin concentrations (mmol/L)
Change in fasting plasma insulin concentrations at week 4 | Baseline and week 4
  Fasting plasma insulin concentrations (mmol/L)
Change in fasting plasma non-esterified fatty acid concentrations at week 12 | Baseline and week 12
  Fasting plasma non-esterified fatty acid concentrations (mmol/L)
Change in fasting plasma non-esterified fatty acid concentrations at week 4 | Baseline and week 4
  Fasting plasma non-esterified fatty acid concentrations (mmol/L)
Change in 7-day mean interstitial glucose concentration at week 12 | Baseline and week 12
  Mean interstitial glucose concentration (mmol/L) measured by continuous glucose monitor over a 7-day period
Change in 7-day standard deviation of interstitial glucose concentration at week 12 | Baseline and Week 12
  Standard deviation of interstitial glucose concentration (mmol/L) measured by continuous glucose monitor over a 7-day period
Change in 7-day coefficient of variation for interstitial glucose concentration at week 12 | Baseline and week 12.
  Coefficient of variation for interstitial glucose concentration (%) measured by continuous glucose monitor over a 7-day period
Change in 7-day mean amplitude of glycaemic excursions for interstitial glucose at week 12 | Baseline and week 12.
  Mean amplitude of glycaemic excursions for interstitial glucose (mmol/L) measured by continuous glucose monitor over a 7-day period

OTHER OUTCOMES:
Change in fasting plasma VLDL-rich triglyceride concentrations at week 12 | Baseline and week 12
  Fasting plasma VLDL-rich triglyceride concentrations (mmol/L)
Change in fasting plasma VLDL-rich triglyceride concentrations at week 4 | Baseline and week 4
  Fasting plasma VLDL-rich triglyceride concentrations (mmol/L)
Change in body mass at week 12 | Baseline and week 12
  Body mass (kg)
Change in body mass at week 4 | Baseline and week 4
  Body mass (kg)
Change in waist-to-hit ratio at week 12 | Baseline and week 12
  Waist-to-hit ratio
Change in waist-to-hit ratio at week 4 | Baseline and week 4
  Waist-to-hit ratio
Change in fat mass at week 12 | Baseline and week 12
  Fat mass determined by dual-energy x-ray absorptiometry (kg)
Change in fat mass at week 4 | Baseline and week 4
  Fat mass determined by dual-energy x-ray absorptiometry (kg)
Change in fat-free mass at week 12 | Baseline and week 12
  Fat-free mass determined by dual-energy x-ray absorptiometry (kg)
Change in fat-free mass at week 4 | Baseline and week 4
  Fat-free mass determined by dual-energy x-ray absorptiometry (kg)
Change in sagittal abdominal diameter at week 12 | Baseline and week 12
  Sagittal abdominal diameter (cm)
Change in sagittal abdominal diameter at week 4 | Baseline and week 4
  Sagittal abdominal diameter (cm)
Change in gut microbiome species richness at week 12 | Baseline and week 12
  Species count in fecal sample (as part of ZOE testing program)

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Health, University of Bath, Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Edinburgh RM, Bradley HE, Abdullah NF, Robinson SL, Chrzanowski-Smith OJ, Walhin JP, Joanisse S, Manolopoulos KN, Philp A, Hengist A, Chabowski A, Brodsky FM, Koumanov F, Betts JA, Thompson D, Wallis GA, Gonzalez JT. Lipid Metabolism Links Nutrient-Exercise Timing to Insulin Sensitivity in Men Classified as Overweight or Obese. J Clin Endocrinol Metab. 2020 Mar 1;105(3):660-76. doi: 10.1210/clinem/dgz104. PMID 31628477
- [Background] Edinburgh RM, Koumanov F, Gonzalez JT. Impact of pre-exercise feeding status on metabolic adaptations to endurance-type exercise training. J Physiol. 2022 Mar;600(6):1327-1338. doi: 10.1113/JP280748. Epub 2021 Jan 27. PMID 33428210